CLINICAL TRIAL: NCT06394154
Title: Validation of the Youth Version of the Alimetry Gut-Brain Wellbeing Survey: A Mental Health Scale for Patients With Chronic Gastroduodenal Symptoms
Brief Title: Validation of a Mental Health Scale for Young People With Chronic Stomach Symptoms
Status: Not yet recruiting | Type: Observational
Sponsor: Greg O'Grady (Other)
Collaborators: University of Auckland, New Zealand (Other)
Responsible Party: Sponsor-Investigator, Greg O'Grady, Professor, University of Auckland, New Zealand
Organization: University of Auckland, New Zealand (Other)
Other Study IDs: AGBW-Y_Val
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Functional Gastrointestinal Disorders; Gastroparesis; Vomiting; Cyclical; Nausea; Vomiting; Rumination Syndrome; Aerophagy; Dyspepsia
MeSH Terms: conditions — Gastrointestinal Diseases; Gastroparesis; Familial cyclic vomiting syndrome; Nausea; Vomiting; Rumination Syndrome; Aerophagy; Dyspepsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to validate the Alimetry® Gut-Brain Wellbeing Survey- Youth Version (AGBW-Y), a mental health scale developed for patients aged 12-17 years with chronic stomach symptoms.

DETAILED DESCRIPTION:
There is currently a lack of validated questionnaires developed to assess mental health within patients with chronic stomach symptoms. Our team has therefore developed and validated a new mental health scale for patients with gastroduodenal symptoms, the Alimetry® Gut-Brain Wellbeing (AGBW) Survey.

However, the AGBW Survey was developed and validated for patients aged 18 years and over. Therefore, the Alimetry® Gut-Brain Wellbeing Survey- Youth Version (AGBW- Y) was developed for use in patients with chronic gastroduodenal symptoms aged 12-17 years. This scale is adapted from the adult AGBW Survey, with more appropriate wording for this age group.

This study will distribute an anonymous, online survey to adolescent patients with chronic gastroduodenal symptoms aged 12-17 years. This survey will ask questions about a patient's general demographics, gastrointestinal symptoms, and mental health in order to assess the validity and reliability of the AGBW-Y.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-17 years
* Able to read and write fluently in English
* Meet the Rome IV criteria and/or have a self-reported previous clinical diagnosis for at least one of the following childhood gastroduodenal DGBIs: gastroparesis, cyclic vomiting syndrome, functional nausea, functional vomiting, rumination syndrome, aerophagia, or functional dyspepsia

Exclusion Criteria:

* Patients with self-induced vomiting
* Patients with an eating disorder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with chronic gastroduodenal symptoms aged 12-17 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Internal Consistency Reliability of the AGBW-Y total score and subscales | Baseline
  Measured via Cronbach's alpha and item-total correlations
Convergent Validity of the AGBW-Y total score and subscales | Baseline
  Pearson's correlation coefficients between the AGBW-Y total score and subscales and the Patient Health Questionnaire for Adolescents (PHQ-A), the Generalized Anxiety Disorder- 7 (GAD-7), the PROMIS Pediatric Psychological Stress Experiences Short Form 8a (PPSE), the Depression Anxiety and Stress Scale Youth Version (DASS-Y), and the Kessler Psychological Distress Scale (K10)
Divergent Validity of the AGBW-Y total score and subscales | Baseline
  Pearson's correlation coefficients between the AGBW-Y total score and subscales and the Big Five Questionnaire for Children (BFQ-C) energy/extraversion subscale and the the Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA)
Concurrent Validity of the AGBW-Y total score and subscales | Baseline
  Pearson's correlation coefficients between the AGBW-Y total score and subscales and the Pediatric Quality of Life Inventory 4.0 (PedsQL)